CLINICAL TRIAL: NCT07363980
Title: Coronary Computed Tomography Angiography In Rheumatoid Arthritis Study
Acronym: COTIRA
Status: Enrolling by invitation | Type: Observational
Sponsor: Ellen Margrethe Hauge (Other)
Collaborators: University of Aarhus (Other); Aarhus University Hospital (Other); Independent Research Fund Denmark (Industry); Alfasigma S.p.A. (Industry); ATACC-RD consortium (Unknown); The Danish Rheumatism Association (Other)
Responsible Party: Sponsor-Investigator, Ellen Margrethe Hauge, Chair professor, University of Aarhus
Organization: University of Aarhus (Other)
Other Study IDs: 1-10-72-85-23
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis; Atherosclerotic Ischemic Disease; Pulmonary Disease; Depressive Disorder; Anxiety Disorders; Cardiovascular and Respiratory Disease; Cardiovascular Biomarkers; Cardiovascular (CV) Risk; Cardiovascular Disease; Cardiovascular Disease (CKD); Cardiovascular Disease (CVD) Risk Factors; COPD (Chronic Obstructive Pulmonary Disease); Pulmonary Diseases or Conditions; Pulmonary Disease, Chronic Obstructive; Depressive and Anxiety Disorders; Interstitial Lung Disease in Patients With Rheumatoid Arthritis; Lung Cancer (Diagnosis)
Keywords: Coronary Computed Tomography Angiography; Pulmonary function tests; Biobank; Faecal microbiome; Patient reported outcomes; Genome sequencing; RNA sequencing; Epigenom sequencing; Coronary Artery Calcium Score; Proteomics; Metabolomics; Lipidomics; Multi-omics; Patient-reported outcomes; Disease Activity Score-28 for Rheumatoid Arthritis; Deep phenotyping; Coronary plaque analysis
MeSH Terms: conditions — Arthritis, Rheumatoid; Lung Diseases; Depressive Disorder; Anxiety Disorders; Respiration Disorders; Cardiovascular Diseases; Pulmonary Disease, Chronic Obstructive; Lung Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Blood biobank
  2. Faeces microbiome biobank
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Coronary Computed Tomography Angiography in Rheumatoid Arthritis study is part of the multinational, prospective, observational Autoimmunity and Atherosclerosis in Rheumatic Diseases cohort (https://atacc-rd.com) that includes comprehensive baseline and follow-up assessments at 3, 5, and 10 years. It comprises a main protocol and several optional modules, including a Cardiac Imaging Module, Biobanking Module, Pulmonary Module, and Anxiety and Depression Module.

The study aims to advance understanding of cardiopulmonary and psychological comorbidities in rheumatoid arthritis, to improve early identification and management, and to enhance insights into underlying disease mechanisms-ultimately refining risk stratification and targeted prevention strategies.

The study includes 4,000 patients with rheumatoid arthritis enrolled through the Cardiac Imaging Module in the main protocol. Participants undergo coronary computed tomography angiography, pulmonary function testing, physical examination, questionnaires, and biobanking, supplemented by genetic, proteomic, metabolomic, and microbiome profiling.

DETAILED DESCRIPTION:
This prospective, observational study follows individuals with rheumatoid arthritis over time to understand how the disease and its treatment relate to cardiovascular, pulmonary, psychological, and biological outcomes. The study collects standardized clinical data from outpatient rheumatology clinics, complemented by advanced imaging, biological sample collection, and linkage to national health registries.

Study Procedures and Visit Schedule Participants are enrolled during routine or ad-hoc outpatient visits. After informed consent, a baseline evaluation is performed, followed by standardized follow-up visits after approximately 3, 5, and 10 years (± 3-6 months).

At baseline, demographic and lifestyle factors (age, sex, education, smoking, alcohol, physical activity, and family history) are recorded together with anthropometric measures (height, weight, waist circumference) and rheumatoid arthritis characteristics (serologic status, disease duration, erosive disease, and disease activity scores). Concomitant diseases and medications are documented, and vital signs and blood pressure are measured.

Patient-reported outcomes include validated questionnaires on quality of life (Short Form 36, version 1), functional ability (Multidimensional Health Assessment Questionnaire), work productivity (Work Productivity and Activity Impairment - General Health), fatigue and pain visual analogue scales, physical activity (International Physical Activity Questionnaire - Short Form), and shortness of breath (University of California, San Diego Shortness of Breath Questionnaire). Laboratory results, including markers of inflammation and metabolic status, are obtained according to routine standards.

Follow-up visits repeat these assessments to evaluate disease activity, lifestyle changes, and incident comorbidities. Events such as hospitalizations, procedures, and deaths are continuously updated through registry linkage, ensuring complete longitudinal follow-up.

Registry Data Sources All participants are linked to national Danish health and administrative registries to enable comprehensive, long-term follow-up. The study integrates data from the National Patient Registry, the Danish Rheumatology Quality Database, the Civil Registration System, the Danish National Causes of Death Registry, the Western Denmark Heart Registry, the Danish Heart Registry, the Danish Stroke Registry, the Danish National Vascular Registry, the Danish National Database of Reimbursed Prescriptions, the Clinical Laboratory Information System, the Register of Laboratory Results for Research, and the Danish Research Institute for Economic Analysis and Modelling. Linkage across these registries allows continuous capture of clinical events, treatments, and vital status, ensuring complete longitudinal follow-up and verification of outcomes recorded during study visits.

Governance The study is governed by an executive steering committee responsible for overall scientific direction, study design, resource allocation, and regulatory compliance. Supporting boards and advisory groups contribute to patient involvement, methodological quality, and international collaboration. Dedicated centers coordinate site operations, biobanking, cardiac imaging, and data analysis to ensure standardized procedures and data integrity across all participating sites.

All procedures are conducted in accordance with Danish and European data-protection regulations, and data are stored and managed in secure systems compliant with the General Data Protection Regulation.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill the ACR/EULAR-2010 criteria for rheumatoid arthritis
* Attending or has attended at least one visit during the last two years in rheumatology outpatient clinic for diagnostic or monitoring purposes related to rheumatoid arthritis
* Age 50-75 years

Exclusion Criteria:

* Diagnosed with overlapping systemic autoimmune diseases other than secondary Sjogren's syndrome
* Active cancer
* Prior coronary atherosclerotic symptoms as defined by myocardial infraction, percutaneous coronary intervention, or coronary artery bypass grafting
* Allergy to radiocontrast agents
* Estimated glomerular filtration rate (eGFR) < 30 mL/min
* BMI > 35 kg/m2
* Persistent atrial fibrillation

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis from rheumatology outpatient clinics across Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2038-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a first occurrence of Major Adverse Cardiovascular Events (MACE) | 3, 5 and 10 years
  1. Cardiovascular death as defined by death from any of the following causes: Ischemic heart disease; Sudden cardiac death; Ventricular tachycardia; Other cardiac arrhythmias; Heart failure; Fatal ischemic stroke; Sudden undefined death; Unwitnessed or unknown cause of death
  2. Hospitalization for non-fatal myocardial infarction, including hospitalization for PCI and CABG
  3. Hospitalization for non-fatal ischemic stroke
Number of participants with a first occurrence of any ischemic cardiovascular events, including MACE | 3, 5 and 10 years
  Hospitalization for cerebrovascular disease (transient ischemic attack). Hospitalization for peripheral vascular disease. Hospitalization for peripheral vascular surgery. Cardiovascular death as defined by death from any of the following causes: Ischemic heart disease; Sudden cardiac death; Ventricular tachycardia; Other cardiac arrhythmias; Heart failure; Fatal ischemic stroke; Sudden undefined death; Unwitnessed or unknown cause of death. Hospitalization for non-fatal myocardial infarction, including hospitalization for PCI and CABG. Hospitalization for non-fatal ischemic stroke
Number of participants with all-cause death (all-cause mortality) | 3, 5 and 10 years
  Death from any cause

SECONDARY OUTCOMES:
Coronary Artery Calcium Score (Agatston score) | Baseline
  Coronary Artery Calcium Score (CACS), Agatston units. Minimum: 0. Maximum: No upper limit. Higher score indicates worse outcome (more coronary artery calcification).
The coronary artery plaque surface extent at baseline evaluated for the percent composition of non-calcified-, mixed-, and calcified plaques | Baseline
  Quantitative plaque measurement
Change in Coronary Artery Calcium Score (Agatston units) from baseline to 3 years | Baseline and 3 years
  Coronary Artery Calcium Score (Agatston score), Agatston units. Change (Δ) in Coronary Artery Calcium Score (CACS) calculated as 3-year CACS minus baseline CACS. Minimum: No lower limit (negative). Maximum: No upper limit (positive). A positive change indicates increasing calcification (worse); a negative change indicates decreasing calcification (better).
The quantitative difference in coronary artery plaque surface extent from baseline to 3 years evaluated for the percent composition of non-calcified-, mixed-, and calcified plaques | Baseline and 3 year
  Quantitative plaque measurement
Number of participants with a occurrence of hospitalization for cerebrovascular disease | 3, 5 and 10 years
  Source of data: patient, record, registry
Number of participants with a first occurrence of hospitalization for non-fatal myocardial infarction | 3, 5 and 10 years
  Source of data: patient, record, registry
Number of participants with a occurrence of hospitalization for non-fatal ischemic stroke | 3, 5 and 10 years
  Source of data: patient, record, registry
Number of participants with a occurrence of hospitalization for peripheral vascular disease | 3, 5 and 10 years
  Source of data: patient, record, registry
Number of participants with a occurrence of hospitalization for peripheral vascular surgery | 3, 5 and 10 years
  Source of data: patient, record, registry
Number of participants with a occurrence of hospitalization for thromboembolic events as defined by deep vein thrombosis and pulmonary embolism | 3, 5 and 10 years
  Source of data: patient, record, registry
Number of participants with a first occurrence of hospitalization for PCI | 3, 5 and 10 years
  Source of data: patient, record, registry
Number of participants with a first occurrence of hospitalization for CABG | 3, 5 and 10 years
  Source of data: patient, record, registry
Number of participants with a first occurrence of treatment for stable angina pectoris | 3, 5 and 10 years
  Source of data: patient, record, registry
Number of participants with a occurrence of treatment for atrial fibrillation and flutter | 3, 5 and 10 years
  Source of data: patient, record, registry
Number of participants with sudden death | 3, 5 and 10 years
  Source of data: record and registry
Number of participants with cardiovascular death | 3, 5 and 10 years
  Source of data: record and registry
Number of participants with a occurrence of treatment for essential hypertension with/without complications | 3, 5 and 10 years
  Source of data: patient, record, registry
Number of participants with a occurrence of treatment for disorders of lipoprotein metabolism and other lipidemias | 3, 5 and 10 years
  Source of data: patient, record, registry
Number of participants with a occurrence of treatment for diabetes mellitus | 3, 5 and 10 years
  Source of data: patient, record, registry
Number of participants with a occurrence of hospitalization for respiratory disease | 3, 5 and 10 years
  Source of data: patient, record, registry
Number of participants with a occurrence of hospitalization or specialist-initiated treatment for interstitial pulmonary diseases | 3, 5 and 10 years
  Source of data: patient, record, registry
Number of participants with a occurrence of hospitalization or specialist-initiated treatment for chronic lower respiratory diseases | 3, 5 and 10 years
  Source of data: patient, record, registry
Number of participants with a occurrence of hospitalization or specialist-initiated treatment for anxiety disorders, including generalized anxiety disorder | 3, 5 and 10 years
  Source of data: patient, record, registry
Number of participants with a occurrence of hospitalization or specialist-initiated treatment for a depressive episode or recurrent major depressive disorder | 3, 5 and 10 years
  Source of data: patient, record, registry
Number of participants with a occurrence of general practitioner-initiated treatment for anxiety disorders | 3, 5 and 10 years
  Source of data: patient, record, registry
Number of participants with a occurrence of general practitioner-initiated treatment for depression | 3, 5 and 10 years
  Source of data: patient, record, registry
Number of participants with a occurrence of referral to a psychologist or psychiatrist | 3, 5 and 10 years
  Source of data: patient, record, registry
Number of participants with a occurrence of infection with Mycobacterium tuberculosis | 3, 5 and 10 years
  Source of data: patient, record, registry
Number of participants with a occurrence of opportunistic infections | 3, 5 and 10 years
  Source of data: patient, record, registry
Number of participants with a occurrence of hospitalization for infections (suspected/confirmed) | 3, 5 and 10 years
  Source of data: patient, record, registry
Proteomics concentrations | Baseline, 3, 5 and 10 years
  Blood sample
Metabolomics concentration | Baseline, 3, 5 and 10 years
  Blood and stool sample
Microbiome profile of stool | Baseline, 3, 5 and 10 years
  Stool sample
Genome-, epigenom-, and RNA sequencing | Baseline, 3, 5 and 10 years
  Blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Ellen-Margrethe Hauge, MD, PhD, Study Chair — Aarhus University Hospital and Aarhus University; Dzenan Masic, MD, PhD, Study Director — Aarhus University Hospital and Aarhus University
Locations (4):
- Denmark (4):
  - Aarhus University Hospital, Aarhus
  - Esbjerg Hospital, Esbjerg
  - Regional Hospital Gødstrup, Herning
  - Silkeborg Regional Hospital, Herning

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the study.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: After completion of the study.
Access Criteria: Individuals who obtain approval from the Danish Ethical Review Authority, the authority responsible for personal data, and the COTIRA Steering Committee will be able to access all PIDs as described above.